CLINICAL TRIAL: NCT00847171
Title: A Safety and Bioactivity Study of Combination Therapy With Trastuzumab, Cyclophosphamide, and an Allogeneic GM-CSF-Secreting Breast Tumor Vaccine for the Treatment of Patients With High Risk/ Metastatic HER-2/Neu- Overexpressing Breast Cancer With No Evidence of Disease
Brief Title: Trastuzumab, Cyclophosphamide, and Vaccine Therapy in Treating Patients With High-Risk or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0885; P30CA006973 (NIH); NA_00021048 (Other: JHM IRB); CDR0000634155 (Other: other)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Cyclophosphamide; Flow Cytometry; Immunoenzyme Techniques; Immunohistochemistry; Biopsy

ARMS (1):
- Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine (Experimental): Participants receive Trastuzumab (T), Cyclophosphamide (CY), and an allogeneic GM-CSF-secreting whole cell breast cancer vaccine
  Interventions: Biological: allogeneic GM-CSF-secreting breast cancer vaccine; Biological: trastuzumab; Drug: cyclophosphamide; Other: flow cytometry; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: biopsy

INTERVENTIONS:
Biological: allogeneic GM-CSF-secreting breast cancer vaccine — Day 0 : Allogeneic GM-CSF-secreting Breast Cancer Vaccine administered as:
  12 intradermal injections of a divided total dose of 5 x108 cells.
Biological: trastuzumab — Patient HAS received prior Trastuzumab within the last two weeks, give Trastuzumab 2 mg/kg weekly on Day -1 for 5 weeks.
  Patient has NOT received Trastuzumab within the last two weeks, give On Cycle 1, Day -1 ONLY, Loading dose 4 mg/kg
  Other Names: Herceptin
Drug: cyclophosphamide — Cyclophosphamide 200mg/m2 IV in NS 100ml over 30 minutes on Day -1 ONLY. Note: there are no dose modifications for Cyclophosphamide.
  Other Names: Cytoxan
Other: flow cytometry — Samples will be analyzed by flow cytometry using Cell Quest software
Other: immunoenzyme technique
Other: immunohistochemistry staining method — Measuring Immune Priming In Vivo By Vaccine Site Biopsies
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy — skin biopsy to be performed on day 3 and day 7 for cycle 1 and 3 only

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vaccines made from gene-modified tumor cells may help the body build an immune response to kill tumor cells. Giving trastuzumab together with cyclophosphamide and vaccine therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving trastuzumab together with cyclophosphamide and vaccine therapy in treating patients with high-risk or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety of allogeneic sargramostim (GM-CSF)-secreting breast cancer vaccine in combination with trastuzumab (Herceptin®) and cyclophosphamide in patients with high-risk or metastatic HER2/neu-overexpressing breast cancer.
* To measure the HER2/neu-specific CD4+ T-cell response by delayed-type hypersensitivity.
* To measure the magnitude of HER2/neu-specific CD8+ T-cell responses by ELISPOT.

Secondary

* To assess the impact of trastuzumab on immune priming in vivo by IHC.
* To measure the impact of cyclophosphamide pretreatment on CD4+CD25+ regulatory T cells by flow cytometry.
* To determine the time to disease progression.

Tertiary

* To develop the tandem tetramer/CD107a cytotoxicity assay for HER2/neu-specific CD8+ T cells.
* To measure novel T-cell responses induced by trastuzumab and cyclophosphamide-modulated vaccination.

OUTLINE: Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes once weekly beginning on day -1 of the first course of vaccination and continuing until the completion of the last course of vaccination. Patients also receive cyclophosphamide IV over 30 minutes on day -1 and allogeneic sargramostim (GM-CSF)-secreting breast cancer vaccine intradermally on day 0. Treatment with cyclophosphamide and the vaccine repeats every 27-42 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive a fourth course of cyclophosphamide and vaccine approximately 6-8 months after the first course.

Patients undergo delayed-type hypersensitivity testing and blood sample collection at baseline and periodically during study for immunologic laboratory studies. Blood samples are analyzed for serum GM-CSF levels by pharmacokinetic studies and for immune monitoring by ELISPOT and flow cytometry. Skin punch biopsies are also performed periodically and analyzed by IHC.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast, meeting one of the following criteria:

  * Metastatic disease
  * High-risk disease, defined as early-stage disease with pathologic involvement of locoregional lymph nodes

    * Patients who are/will be receiving standard adjuvant trastuzumab [Herceptin®] for high-risk disease will participate in this study during the single-agent trastuzumab portion of their therapy
* No clinical or radiographical evidence of active disease
* Not eligible for therapy of known curative potential for metastatic breast cancer
* HER2/neu-overexpressing disease, defined as HER2/neu positive by IHC 3+ staining or by FISH+ amplification
* Stable CNS disease allowed provided it has been adequately treated and is not under active treatment
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* ANC > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Serum creatinine < 2.0 mg/dL
* Serum bilirubin ≤ 2.0 mg/dL (unless elevation is due to known Gilbert's syndrome)
* AST/ALT ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Cardiac ejection fraction normal by MUGA OR ≥ 45% by ECHO
* No other malignancies within the past 5 years, except for carcinoma in situ of the cervix, superficial nonmelanoma skin cancer, or superficial bladder cancer
* No prior or currently active autoimmune disease* requiring management with systemic immunosuppression, including any of the following:

  * Inflammatory bowel disease
  * Systemic vasculitis
  * Scleroderma
  * Psoriasis
  * Multiple sclerosis
  * Hemolytic anemia or immune-mediated thrombocytopenia
  * Rheumatoid arthritis
  * Systemic lupus erythematosus
  * Sjögren syndrome
  * Sarcoidosis
  * Other rheumatologic disease
* No symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest
* HIV-negative
* No evidence of active acute or chronic infection
* No uncontrolled medical problems
* No active major medical or psychosocial problems that could be complicated by study participation
* No corn allergy
* No known severe hypersensitivity to trastuzumab (except for mild to moderate infusion reactions that are easily managed and do not recur) NOTE: *Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids allowed

PRIOR CONCURRENT THERAPY:

* Any number of prior chemotherapy regimens for metastatic breast cancer allowed
* Prior or concurrent trastuzumab in the adjuvant or metastatic setting allowed
* More than 28 days since prior and no concurrent systemic oral steroids

  * Topical, ocular, or nasal steroids allowed
* More than 28 days since prior and no concurrent chemotherapy, radiotherapy, or biologic therapy (except trastuzumab)
* More than 28 days since prior and no concurrent participation in another investigational clinical trial involving a new drug
* Concurrent endocrine therapy or bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leisha A. Emens, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine: Patients receive Trastuzumab (T), Cyclophosphamide (CY), and an allogeneic GM-CSF-secreting whole cell breast cancer vaccine
Period: Overall Study
Arm/Group | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 47 [34 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Number of Participants Experiencing Toxicity
Description: Safety as assessed by number of participants who experienced drug-related local and systemic toxicity, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v3.0) in response to CY-modulated immunization with a novel breast cancer vaccine in the setting of weekly Trastuzumab therapy.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Groups:
- Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine: All patients receive weekly Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
Arm/Group | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
Number analyzed (Participants) | 20
Participants
  Patients with drug-related toxicity | 20
  Patients with grade 3+ drug-related toxicity | 0
  Patients with serious drug-related toxicity | 0

2. Primary Outcome: Number of Participants With Immunologic Response as Determined by Delayed-type Hypersensitivity (DTH) Response to HER2/Neu-derived Peptides
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
Number analyzed (Participants) | 20
Participants
  DTH-positive at baseline | 12
  Increased DTH from baseline | 11
  Converted from DTH-negative to DTH-positive | 5

3. Secondary Outcome: Clinical Benefit as Assessed by Number of Participants With Progression-free Survival
Description: Number of participants without evidence of disease progression.
Time Frame: 4 years
Population: Only 13/20 participants had early stage disease, and 7/20 participants had a history of metastatic disease at the start of the study. All participants were assigned to the same treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
Number analyzed (Participants) | 20
Participants
  Patients with early stage disease: number analyzed (Participants) | 13
  Patients with early stage disease | 12
  Patients with metastatic disease: number analyzed (Participants) | 7
  Patients with metastatic disease | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected at weekly time points after each vaccine administration for the duration of the study, an average of 7 months.
Arm/Group | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Cyclophosphamide, and a Breast Tumor Vaccine (N=20)
Erythema/swelling of vaccine sites (Skin and subcutaneous tissue disorders) | 20
Pain/soreness/tenderness of vaccine sites (Skin and subcutaneous tissue disorders) | 20
Pruritus of vaccine sites (Skin and subcutaneous tissue disorders) | 20
Blister at vaccine site (Skin and subcutaneous tissue disorders) | 16
Dry skin at vaccine site (Skin and subcutaneous tissue disorders) | 1
Ecchymosis at vaccine site (Skin and subcutaneous tissue disorders) | 6
Eczema at vaccine site (Skin and subcutaneous tissue disorders) | 1
Edema at vaccine site (Skin and subcutaneous tissue disorders) | 1
Hives at vaccine site (Skin and subcutaneous tissue disorders) | 2
Hyperpigmentation at vaccine site (Skin and subcutaneous tissue disorders) | 1
Rash at vaccine site (Skin and subcutaneous tissue disorders) | 2
Warmth at vaccine site (Skin and subcutaneous tissue disorders) | 14
Anorexia (Gastrointestinal disorders) | 5
Arthralgia (General disorders) | 9
Blisters (Skin and subcutaneous tissue disorders) | 2
Chills (General disorders) | 10
Constipation (Gastrointestinal disorders) | 1
Cramps (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 10
Fever (General disorders) | 7
Flu-like symptoms (General disorders) | 3
Headache (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 4
Malaise (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 4
Pain, bone (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Sweats (General disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes